CLINICAL TRIAL: NCT03337568
Title: Allogeneic HCT From Donor-sources of Matched-sibling, Matched-unrelated, or Haploidentical-family Donors Using Uniform Conditioning Regimen of Busulfan, Fludarabine, and Antithymocyte Globulin for AML in Remission - an Observational Study
Brief Title: Allogeneic HCT Using Uniform Conditioning Regimen Regardless of Donors (MS, MU, or HF) for AML in Remission
Acronym: AML_AlloHCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Research Institute of Bioscience & Biotechnology (Other Government)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, MD, Professor, Asan Medical Center
Other Study IDs: 2017-0204
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML CR; allogeneic hematopoietic cell transplantation; busulfan; fludarabine; ATG
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: allogeneic hematopoietic cell transplantation — perform allogeneic hematopoietic cell transplantation (HCT) using conditioning regimen of busulfan, fludarabine, and antithymocyte globulin

SUMMARY:
The purpose of this study is to evaluate the effect of various clinical variables including HLA-disparity and NK cell-related variables, upon outcomes of allogeneic hematopoietic cell transplantation (HCT) using uniform conditioning regimen including busulfan, fludarabine, and antithymocyte globulin (ATG) in patients with acute myeloid leukemia (AML) in the first complete remission (CR). The donors for allogeneic HCT include HLA-matched siblings, matched unrelated donors, and haploidentical family donors.

Therefore, the endpoints of the study are engraftment, secondary graft failure, acute and chronic graft-versus-host disease (GVHD), immune recovery, infections, leukemia recurrence, non-relapse mortality, and relapse-free (RFS) and overall survival (OS) of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-promyelocytic AML (intermediate-risk or high-risk diseases by NCCN guideline 2016) in the first CR
* Patients should be 16 years of age or more and 75 years of age or less
* The performance status of the patients should be 70 or over by Karnofsky performance scale
* Patients should have adequate hepatic function (bilirubin less than 2.0 mg/dl, AST less than three times the upper normal limit)
* Patients should have adequate renal function (creatinine less than 2.0 mg/dl)
* Patients should have adequate cardiac function (ejection fraction > 40% on MUGA scan)
* Patients and stem cell donors must sign informed consent
* For hematopoietic cell donor, if a patient has an HLA-matched sibling (65 years or younger), that sibling will be a cell donor. If a patient does not have an HLA-matched sibling but an HLA-A, B, C, DRB1 7-8/8 matched unrelated donor, the unrelated donor will be a cell donor. If a patient has neither HLA-matched sibling nor unrelated donor, an HLA-haploidentical familial donor will be a cell donor.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a single center, observational study in a patient population with non-promyelocytic AML who have achieved complete remission after induction chemotherapy. The patients will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
leukemia recurrence | from HCT (day of donor cell infusion) to leukemia recurrence at 2 years after HCT
  reappearance of blast >5% in bone marrow; reappearance of leukemia blast in extramedullary sites
engraftment | from HCT to neutrophil count over >500/uL at 30 days after HCT
  recovery of absolute neutrophil count over >500/uL
GVHD, acute and chronic | from HCT to the occurrence of GVHD at 2 years after HCT
  occurrence of acute or chronic GVHD after HCT
Non-relapse mortality | from HCT to the occurrence of death without leukemia recurrence at 2 years after HCT
  occurrence of death without leukemia recurrence

SECONDARY OUTCOMES:
relapse free survival | from HCT to last the follow-up, leukemia recurrence, or death at 2 years after HCT
  survival without leukemia recurrence/death
overall survival | from HCT to the last follow-up or death at 2 years after HCT
  survival regardless of leukemia recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo-Hyung Lee, MD, Principal Investigator — University of Ulsan, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KH, Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Hwang HJ, Jung AR, Kim SH, Yun SC, Shin HJ. Reduced-intensity conditioning therapy with busulfan, fludarabine, and antithymocyte globulin for HLA-haploidentical hematopoietic cell transplantation in acute leukemia and myelodysplastic syndrome. Blood. 2011 Sep 1;118(9):2609-17. doi: 10.1182/blood-2011-02-339838. Epub 2011 Jun 28. PMID 21715313
- [Result] Lee KH, Lee JH, Lee JH, Kim DY, Park HS, Choi EJ, Ko SH, Seol M, Lee YS, Kang YA, Jeon M, Baek S, Kang YL, Kim SH, Yun SC, Kim H, Jo JC, Choi Y, Joo YD, Lim SN. Reduced-Intensity Conditioning with Busulfan, Fludarabine, and Antithymocyte Globulin for Hematopoietic Cell Transplantation from Unrelated or Haploidentical Family Donors in Patients with Acute Myeloid Leukemia in Remission. Biol Blood Marrow Transplant. 2017 Sep;23(9):1555-1566. doi: 10.1016/j.bbmt.2017.05.025. Epub 2017 May 25. PMID 28552421
- [Derived] Choi Y, Choi EJ, Park HS, Lee JH, Lee JH, Lee YS, Kang YA, Jeon M, Woo JM, Kang H, Baek S, Kim SM, Bong CE, Lee KH. A uniform conditioning regimen of busulfan, fludarabine, and antithymocyte globulin for allogeneic haematopoietic cell transplantation from haploidentical family, matched sibling, or unrelated donors-A single-centre, prospective, explorative study. Br J Haematol. 2023 Mar;200(5):608-621. doi: 10.1111/bjh.18550. Epub 2022 Nov 12. PMID 36370064